CLINICAL TRIAL: NCT03145155
Title: Integrating Services for Noncommunicable Diseases in Continuum of Care for Mothers and Children: a Cluster Randomized Control Trial in Myanmar
Brief Title: Integrating Services for Noncommunicable Diseases in Continuum of Care for Mothers and Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokyo University (Other)
Collaborators: Japan Agency for Medical Research and Development (Other Government)
Responsible Party: Principal Investigator, Moe Moe Thandar, PhD candidate, Department of Community and Global Health, School of International Health, Graduate School of Medicine, Tokyo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 11498
Record Dates: First submitted 2017-04-20; First posted 2017-05-09 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Continuum of Care; Noncommunicable Diseases
Keywords: continuum of care; maternal; newborn; child health; noncommunicable diseases
MeSH Terms: conditions — Noncommunicable Diseases | interventions — Continuity of Patient Care

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Pregnant women in intervention arm will receive CoC card and health education on CoC in maternal, newborn and child health (MNCH), NCD and nutrition. The CoC card will include CoC services from first antenatal care(ANC) to last postnatal care(PNC) including four ANC, skilled birth attendance (SBA) and four PNC and essential services. Pregnant women will get stickers if they receive above services. Health education will be given three times during pregnancy and one time during postpartum period.
  Interventions: Behavioral: Integrating services for noncommunicable diseases in continuum of care for mothers and children
- Control (Placebo Comparator): Pregnant women in control arm will receive ordinary health education on pregnancy care
  Interventions: Behavioral: Ordinary health education for pregnant women

INTERVENTIONS:
Behavioral: Integrating services for noncommunicable diseases in continuum of care for mothers and children — The intervention package will comprise of two components, (1) utilization of CoC card and (2) health education on CoC in maternal, newborn and child health (MNCH), NCD and nutrition. The CoC card will be distributed to mothers by midwives at the time of receiving ANC. The CoC card includes CoC services from first antenatal care(ANC) to last postnatal care(PNC) including four ANC, skilled birth attendance (SBA) and four PNC and essential services. Pregnant women will get stickers if they receive above services. Health education will be given by Public Health Supervisors 2 at the health facilities. Health education will be given three times during pregnancy and one time during postpartum period with pamphlets and posters.
  Arms: Intervention
Behavioral: Ordinary health education for pregnant women — The ordinary health education intervention will cover schedule for ANC, delivery and PNC; danger signs; birth preparedness and nutrition. Health education will be given three times during pregnancy and one time during postpartum period with pamphlets and posters.
  Arms: Control

SUMMARY:
The objectives of this cluster randomized control trial are to examine the effect of combined intervention of the utilization of continuum of care (CoC) card and health education on the completion of CoC services among mothers and to examine the effect of health education on NCDs and nutrition on mothers' knowledge on NCDs and nutrition in Myanmar. Pregnant women between 12-20 weeks of pregnancy will be recruited and assigned into intervention arm (n=600) and control arm (n=600). The intervention package will comprise of two components, (1) utilization of CoC card and (2) health education on CoC in maternal, newborn and child health (MNCH), NCD and nutrition. The CoC card will include CoC services from first antenatal care(ANC) to last postnatal care(PNC) including four ANC, skilled birth attendance (SBA) and four PNC and essential services. Pregnant women will get stickers if they receive above services. Health education will be given three times during pregnancy and one time during postpartum period. Health education will include importance of continuous uptake of MNCH services, NCDs and nutrition. The outcomes are proportion of completion of CoC services and knowledge on NCDs and nutrition.

DETAILED DESCRIPTION:
Antenatal care (ANC) is an important entry point for subsequent use of delivery and postnatal care (PNC) services. When women receive high-quality ANC, they will have skilled birth attendant (SBA) at delivery and continue to receive postnatal care. Continuous uptake of above services is necessary to improve health and well being of maternal, newborn and child health (MNCH). Moreover, the continuum of Care (CoC) offers the critical entry point for women and children for preventive care and health promotion on noncommunicable diseases (NCDs). ANC and PNC visits for women and a series of immunization for children are crucial opportunities to provide integrated services of NCDs. The integration of NCDs prevention and control programs in MNCH services would empower women to control NCDs in their families. However, no study has examined the effect of antenatal health education on CoC on completion of CoC among mothers in Myanmar. In addition, no study has examined the effect of antenatal health education on NCDs and nutrition on knowledge on NCDs and nutrition, and on maternal complications among mothers in Myanmar.

A cluster randomized controlled trial will be done among pregnant women living in study area. The unit of randomization in this study will be "rural health center (RHC)". In each RHC, there are at least four Sub-centers (SCs). RHC including SCs will be considered as one cluster. The investigators will advocate midwives (MW) on the CoC in MNCH and introduce the CoC card. The investigators will also recruit and train Public Health Supervisors 2 (PHS2) in each cluster to provide health education to pregnant women on CoC in MNCH, NCDs and nutrition.

We will conduct the study in three townships (Pantanaw, Inapu, Wakema,) in Ayeyarwaddy region, Myanmar from May 2017 to March 2018. There are a total of 22 health facilities. Out of 22 health facilities in 3 townships, eleven will be allocated into intervention arm and another 11 into control arm. An analyst, who will not be a primary member of the study team, will conduct randomization of clusters using computer-generated random sequences. Estimated sample size of 1200 pregnant women will be recruited, roughly 400 pregnant women in each township. The investigators estimate that about 28 women will seek ANC within one month in each cluster. In total of 22 clusters, the investigators estimate 600 women will seek ANC within one month; therefore, the enrollment period will take two months to get the targeted sample size of 1,200 pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women
* 18 years and above
* between 12-20 weeks of pregnancy at the time of first ANC

Exclusion Criteria:

* younger than 18 years
* first ANC before 12 weeks or after 20 weeks
* mentally ill
* migrant and mobile people

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 630 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Completion of continuum of care | 3 months after delivery
  Proportion of mothers who complete four antenatal care visits, skilled birth attendance and four postnatal care visits

SECONDARY OUTCOMES:
Change in knowledge on NCDs and nutrition | Baseline and 3 months after delivery
  Proportion of mothers who change their knowledge related to NCDs after health education on NCDs and nutrition

CONTACTS AND LOCATIONS:
Overall Officials: Moe Moe Thandar, Principal Investigator — Tokyo University
Locations (1):
- University of Tokyo, Bunkyō, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Raw dataset with unique ID
Supporting Information: Study Protocol
Time Frame: 29 January 2026 to 31 Jauary 2030
URL: https://doi.org/10.5281/zenodo.18416868

REFERENCES:
- [Background] Wang W, Hong R. Levels and determinants of continuum of care for maternal and newborn health in Cambodia-evidence from a population-based survey. BMC Pregnancy Childbirth. 2015 Mar 19;15:62. doi: 10.1186/s12884-015-0497-0. PMID 25885596
- [Background] Kerber KJ, de Graft-Johnson JE, Bhutta ZA, Okong P, Starrs A, Lawn JE. Continuum of care for maternal, newborn, and child health: from slogan to service delivery. Lancet. 2007 Oct 13;370(9595):1358-69. doi: 10.1016/S0140-6736(07)61578-5. PMID 17933651
- [Background] Tinker A, ten Hoope-Bender P, Azfar S, Bustreo F, Bell R. A continuum of care to save newborn lives. Lancet. 2005 Mar 5-11;365(9462):822-5. doi: 10.1016/S0140-6736(05)71016-3. No abstract available. PMID 15752509
- [Background] Yeji F, Shibanuma A, Oduro A, Debpuur C, Kikuchi K, Owusu-Agei S, Gyapong M, Okawa S, Ansah E, Asare GQ, Nanishi K, Williams J, Addei S, Tawiah C, Yasuoka J, Enuameh Y, Sakeah E, Wontuo P, Jimba M, Hodgson A; Ghana EMBRACE Implementation Research Project Team. Continuum of Care in a Maternal, Newborn and Child Health Program in Ghana: Low Completion Rate and Multiple Obstacle Factors. PLoS One. 2015 Dec 9;10(12):e0142849. doi: 10.1371/journal.pone.0142849. eCollection 2015. PMID 26650388
- [Background] Gounder CR, Chaisson RE. A diagonal approach to building primary healthcare systems in resource-limited settings: women-centred integration of HIV/AIDS, tuberculosis, malaria, MCH and NCD initiatives. Trop Med Int Health. 2012 Dec;17(12):1426-31. doi: 10.1111/j.1365-3156.2012.03100.x. Epub 2012 Nov 1. No abstract available. PMID 23113824
- [Background] Kapur A. Links between maternal health and NCDs. Best Pract Res Clin Obstet Gynaecol. 2015 Jan;29(1):32-42. doi: 10.1016/j.bpobgyn.2014.04.016. Epub 2014 Aug 17. PMID 25199858
- [Background] Say L, Chou D, Gemmill A, Tuncalp O, Moller AB, Daniels J, Gulmezoglu AM, Temmerman M, Alkema L. Global causes of maternal death: a WHO systematic analysis. Lancet Glob Health. 2014 Jun;2(6):e323-33. doi: 10.1016/S2214-109X(14)70227-X. Epub 2014 May 5. PMID 25103301